CLINICAL TRIAL: NCT07356453
Title: A Phase 1 Study of PARG Inhibitor FORX-428 in Patients With Advanced Solid Tumors With BRCA1/2 Mutations or Other DDR Deficiencies or High Replication Stress.
Brief Title: A Study of PARG Inhibitor FORX-428 in Patients With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: FoRx Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FORX-428-101
Record Dates: First submitted 2025-12-23; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- First-in-human single-arm, open-label, multicenter Phase 1 dose escalation/expansion cohort study. (Experimental): FORX 428 dose levels planned in the study: Dose Level 1: 30 mg, daily; Dose Level 2: 60 mg, daily; Dose Level 3: 120 mg, daily; Dose Level 4: 200 mg, daily; Dose Level 5: 300 mg, daily; and Dose Level 6: 400 mg, daily. Following the selection of the Recommended Cohort Expansion Dose during Part 1 of the study, new patients will be included in 3 cohorts, with simultaneous parallel enrollment. Patients will be allowed to continue to receive FORX-428 monotherapy until disease progression or unacceptable toxicity. Part 2 will include approximately up to 29 evaluable patients in each expansion cohort as determined by the Simon's optimal 2-stage design. In Stage 1 of each cohort of Part 2, a total number of 10 patients will be accrued. If there are 1 or fewer responses by RECIST version 1.1 among these 10 patients, further enrollment in that cohort will be halted for futility. Otherwise, an additional 19 patients will be accrued per cohort in Stage 2 of Part 2.
  Interventions: Drug: FORX-428

INTERVENTIONS:
Drug: FORX-428 — FORX-428 drug product is formulated as immediate release tablets for oral administration in 3 dosage strengths containing 10 mg, 50 mg, and 100 mg FORX-428 drug substance.

SUMMARY:
The goal of this interventional study is to evaluate the safety and tolerability of escalating doses of FORX-48 as monotherapy in patients with select advanced solid tumors with BRCA1/2 mutations or other DDR deficiencies or high replication stress, and to determine the maximum tolerated dose (MTD) and Recommended Cohort Expansion Dose (RCED) of FORX-428 as monotherapy.

DETAILED DESCRIPTION:
The primary objective of the Expansion cohorts (Part 2) of this study is to evaluate the preliminary anti-tumor activity of FORX-428 as monotherapy.

Secondary Outcome Measures:

The secondary objectives of Part 1 of this study are the following:

* To evaluate the preliminary anti-tumor activity of FORX-428 as monotherapy;
* To evaluate the PK profile of FORX-428 when administered as monotherapy; and
* To evaluate a FORX-428-induced effect on heart rate-corrected QT interval (QTc).

The secondary objectives of Part 2 of this study are the following:

* To evaluate the safety and tolerability of FORX-428 as monotherapy; and
* To evaluate the PK profile of FORX-428 when administered as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be >/=18 years of age at time of signing informed consent;
2. Patient has histologically and/or cytologically confirmed diagnosis of advanced or metastatic selected solid tumors.
3. Patient must have progressed on at least 1 prior line of therapy in the advanced or metastatic setting that is considered an appropriate standard of care. In general, if maintenance therapy is part of the standard of care, it should be considered as part of the "1 prior line of therapy in the advanced or metastatic setting" requirement;
4. Patient must fulfill genomic selection criteria: prior available documented evidence in tissue or blood (circulating tumor DNA [ctDNA]) of the genetic alterations indicated below. The Sponsor Medical Monitor or delegate must confirm eligibility based on the reported genomic alteration and applicable assay cut off criteria prior to patient enrollment.

   • Patients with BRCA1/2 mutations (germline or somatic, pathogenic or likely pathogenic) and other mutations signifying HR deficiency or high replication stress.

   • For Dose Expansion: Tumor types for Dose Expansion cohorts include a subset of tumors specified in Inclusion Criterion 3 as follows: i) Cohort 1: Advanced or metastatic breast cancer independent of hormone receptor status and documented evidence of prior treatment with a locally approved PARP inhibitor(s); ii) Cohort 2: Advanced or metastatic ovarian cancer with prior available documented evidence in tissue or blood (ctDNA) of specific genomic abnormalities.

   iii) Cohort 3: Advanced or metastatic breast cancer with prior available documented evidence in tissue or blood (ctDNA) of specific genomic abnormalities.

   Note: Diagnostic genetic testing for Dose Escalation/backfilling and Dose Expansion cohorts must meet the following requirements:

   • United States (US): Testing must have been performed using a College of American Pathologists/Clinical Laboratory Improvement Amendments (CAP/CLIA)-certified laboratory developed test (LDT) or a Food and Drug Administration (FDA)-approved diagnostic test.
5. Patient has measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 at Clinical Screening; Note: Tumor lesions situated in a previously irradiated or otherwise locally treated area will be considered measurable provided that there has been clear imaging-based progression of the lesion since the time of local treatment.
6. Patient has adequate bone marrow and organ function, defined by the following laboratory results obtained within 14 days before first dose of study drug:

   * Platelet count >/=100 × 10^9/L (>/=100,000/μL) (absence of platelet transfusion within 1 week);
   * Hemoglobin >/=90 g/L (>/=5.6 mmol/L) (absence of red blood cell transfusion within 2 weeks);
   * Absolute neutrophil count >/=1.5 × 10^9/L (>/=1500/μL) (absence of growth factors within 2 weeks);
   * Aspartate aminotransferase and alanine aminotransferase </=2.5 × upper limit normal (ULN) or </=5 × ULN for patients with liver metastases;
   * Total bilirubin </=1.5 × ULN, or </=3.0 × ULN for patients with liver metastases or Gilbert's syndrome;
   * Estimated glomerular filtration rate >/=60 mL/min calculated by the 2021 Chronic Kidney Disease Epidemiology Collaboration Equation; and
   * Adequate coagulation test results defined by activated partial thromboplastin time </=1.5 × ULN, international normalized ratio (INR) </=2.0 with the exception of INR 2 to 3 acceptable for patients on warfarin anticoagulation or direct oral anticoagulants.
7. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2 with >/=3 months of life expectancy for Dose Escalation cohorts, and an ECOG PS of 0 to 1 with >/=3 months of life expectancy for backfilling and Dose Expansion cohorts;
8. Patient is able to swallow tablets and has no gastrointestinal conditions affecting absorption.

Exclusion Criteria:

1. Patient has received anti-cancer treatment or an investigational agent </=14 days or 5 half-lives prior to first dose, whichever is shorter, or patient has received immunotherapy </=28 days prior to first dose; Note: Localized radiotherapy given with palliative intent is allowed and should be completed 1 week or more before receiving the first dose of FORX-428. It may also be allowed after the dose-limiting toxicity (DLT) Observation Period, pending discussion with the Sponsor Medical Monitor or delegate and their approval.
2. Patient has had previous exposure to a PARG inhibitor;
3. Patient has a history of other malignancy diagnosed </=5 years prior to consent, except for any locally occurring cancer that has been treated with curative intent with no evidence of disease for >2 years at the time of consent and includes the following: completely resected cervical carcinoma in situ, basal or squamous cell skin cancer, ductal carcinoma in situ, superficial bladder cancer, or early-stage prostate cancer which has been adequately treated;
4. Patient has had major surgery within 30 days prior to first dose of study drug (with exceptions further defined in the protocol), or anticipation of major surgery during study treatment;
5. Patient has impaired cardiovascular function or clinically significant cardiovascular disease as further stipulated in the protocol;
6. Patient has uncontrolled HIV or hepatitis C infection;
7. Patient has known metastatic central nervous system malignant disease or leptomeningeal disease; Note: Patients previously treated for brain metastasis who are asymptomatic, receiving </=10 mg/day prednisone equivalent, not requiring anti-epileptic therapy, and without evidence of radiological progression for at least 4 weeks are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase: Incidence of Dose-Limiting Toxicities (DLTs) | 1 year.
Dose Escalation Phase: Incidence of treatment-emergent serious adverse events (TESAEs) | 1 year.
Dose Escalation Phase: Incidence and severity of Treatment-emergent adverse event (TEAEs) and laboratory abnormalities | 1 year.
  Adverse events will be recorded and severity graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Dose Escalation Phase: Incidence of treatment discontinuations and treatment modifications due to adverse events (AEs) and laboratory abnormalities | 1 year.
Dose Escalation Phase: Change in vital signs measurements, clinical laboratory assessment, 12-lead electrocardiograms (ECGs), physical examinations (including Eastern Cooperative Oncology Group [ECOG] Performance Status [PS]), and urinalyses | 1 year.
Dose Escalation Phase: Establishing the Maximum Tolerated Dose (MTD) and Recommended Cohort Expansion Dose (RCED) of FORX-428 administered as monotherapy | 1 year.
Dose Expansion Phase: Tumor response: Best Overall Response (BOR) | 1 year.
  BOR will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Dose Expansion Phase: Tumor response: Overall Response Rate (ORR) | 1 year.
  ORR will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Dose Expansion Phase: Tumor response: Disease Control Rate (DCR) | 1 year.
  DCR will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Dose Expansion Phase: Tumor response: Progression-free Survival (PFS) | 1 year.
  PFS will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Dose Expansion Phase: Tumor response: Overall Survival (OS) | 1 year.
  OS will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Dose Escalation Phase: Tumor response: Overall Response Rate (ORR) | 1 year.
  ORR will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Dose Escalation Phase: Tumor response: Best Overall Response (BOR) | 1 year.
  BOR will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Dose Escalation Phase: Tumor response: Disease Control Rate (DCR) | 1 year.
  DCR will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Dose Escalation Phase: Tumor response: best change in tumor size | 1 year.
  Best change in tumor size will be measured according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Dose Escalation Phase: Tumor response: Progression-free Survival (PFS) | 1 year.
Dose Escalation Phase: Tumor response: Overall Survival (OS) | 1 year.
Dose Escalation Phase: Determination of plasma concentrations of FORX-428 | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma (maximum plasma concentration [Cmax]) | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma (time to maximum concentration [Tmax]) | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma area under the plasma concentration curve [AUC] from time 0 to the time of last quantifiable plasma concentration [AUC0 t] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma area under the plasma concentration curve [AUC] from time 0 to time τ [AUCτ] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma area under the plasma concentration curve [AUC] from time 0 to infinity [AUC∞] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma apparent first-order terminal elimination rate constant [λz] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma terminal elimination half-life [t½] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma mean residence time (MRT) | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma apparent clearance [CL/F] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma apparent volume of distribution [Vz/F] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma peak to trough fluctuation [PTF] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma ratio of AUC [RAUC] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma ratio of Cmax [RCmax] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma average plasma concentration at steady state [Css av] | 1 year.
Dose Escalation Phase: PK parameters of FORX-428 when administered as monotherapy in plasma trough plasma concentration [Ctrough] | 1 year.
Dose Escalation Phase: Determination of concentration-QTc | 1 year.
Dose Expansion Phase: Incidence of treatment-emergent serious adverse events (TESAEs) and laboratory abnormalities | 1 year.
  Adverse events will be recorded and severity graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Dose Expansion Phase: Incidence of treatment discontinuations and treatment modifications due to AEs and laboratory abnormalities | 1 year.
Dose Expansion Phase: Change in vital signs measurements, clinical laboratory assessment, 12-lead electrocardiograms (ECGs), physical examinations (including Eastern Cooperative Oncology Group [ECOG] Performance Status [PS]), and urinalyses | 1 year.
Dose Expansion Phase: PK parameters of FORX-428 when administered as monotherapy in plasma (Cmax, tmax, AUC0 t, AUCτ, AUC∞, λz, t½, MRT, CL/F, Vz/F, PTF, RAUC, RCmax, Css av, and Ctrough, as applicable) | 1 year.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Stanford University Medical Center, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - START - Midwest, Grand Rapids, Michigan
  - Washington University St. Louis, St Louis, Missouri
  - Knight Cancer Institute, Portland, Oregon
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - START - San Antonio, San Antonio, Texas
  - NEXT - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No